CLINICAL TRIAL: NCT02272959
Title: Attention Bias Modification Treatment for Children With Anxiety Disorders Who do Not Respond to Cognitive Behavioral Therapy: A Randomized Controlled Trial
Brief Title: Attention Bias Modification Treatment (ABMT) for Anxiety Disorders in Youth Who do Not Respond to CBT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yair Bar-Haim (Other)
Collaborators: United States - Israel Binational Science Foundation (Other); Schneider Children's Hospital (Other); Sheba Medical Center (Other Government)
Responsible Party: Sponsor-Investigator, Yair Bar-Haim, Professor of Psychology and Neuroscience, Head School of Psychological Sciences, Tel Aviv University
Organization: Tel Aviv University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: loe140498ctil
Record Dates: First submitted 2014-10-21; First posted 2014-10-23 (Estimated); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Anxiety Disorders
Keywords: Anxiety/Anxiety disorders, Clinical trials, treatment, cognition, computer/Internet technology
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Attention Bias Modification treatment (ABMT) (Experimental): Attention training via repeated trials of a dot-probe task intended to direct attention away from threat stimuli using threat and neutral stimuli.
  Interventions: Behavioral: Attention bias modification treatment (ABMT)
- Placebo Group (Placebo Comparator): Attention training via repeated trials of a dot-probe task not intended to change threat-related attention patterns using only neutral stimuli.
  Interventions: Behavioral: Attention Control Condition

INTERVENTIONS:
Behavioral: Attention bias modification treatment (ABMT) — Attention training using a computerized spatial attention task (dot-probe) modified to alter threat-related attention patterns using threat and neutral stimuli.
  Arms: Attention Bias Modification treatment (ABMT)
Behavioral: Attention Control Condition — Attention training using a computerized spatial attention task (dot-probe) not intended to alter threat-related attention patterns using only neutral stimuli.
  Arms: Placebo Group

SUMMARY:
First-line psychosocial treatments for anxiety disorders in children are largely exposure-based cognitive behavioral therapies (CBTs). Despite strong evidence supporting CBT's efficacy, for up to 50% of youth patients, symptoms of anxiety persist after a full course of treatment. What are the treatment options for these youth? Unfortunately, there is not a single empirical study in the youth anxiety treatment literature that has systematically examined treatment augmentation for youth who fail to respond to CBT. Empirical efforts to address this issue are important because youth who do not respond to CBT continue to suffer emotional distress and impairment associated with anxiety disorders. This study will address this gap via double-blind randomized controlled trial of Attention Bias Modification Treatment (ABMT) for anxious 10-18 year-olds who did not respond to standard CBT. Attention biases in threat processing have been assigned a prominent role in the etiology and maintenance of anxiety disorders. ABMT utilizes computer-based protocols to implicitly modify biased attentional patterns in anxious patients. Here, participants will be CBT non-responders who will be assessed by using clinical interviews and parent- and self-rated questionnaires before and after eight sessions of ABMT or placebo control, and again at an eight-week follow-up. We expect to see reduction in anxiety symptoms in the Attention Bias Modification Treatment (ABMT) group relative to the placebo control group. We also expect the findings to inform pathways to treatments for anxious children who do not respond to current standard first-line therapy, and to provide initial information on mechanisms of ABMT efficacy.

ELIGIBILITY:
Inclusion Criteria:

To be included all youth must:

1. have received a full course of CBT and were deemed treatment non-responders.
2. they must still have a primary diagnosis of GAD, SOP, or SAD.
3. if they have comorbid attention deficit hyperactivity disorder (ADHD) or depressive disorders, it must be treated with medication and stable.
4. if they have tics or impulse control problems, those problems must be treated with medication and stable and cause minimal or no impairment.

Exclusion Criteria: To be excluded youth must:

1. meet diagnostic criteria for Organic Mental Disorders, Psychotic Disorders, Pervasive Developmental Disorders, or Mental Retardation.
2. show high likelihood of hurting themselves or others.
3. have not been living with a primary caregiver who is legally able to give consent for the child's participation.
4. be a victim of previously undisclosed abuse requiring investigation or ongoing supervision.
5. be involved currently in another psychosocial treatment.
6. have a serious vision problem that is not corrected with prescription lenses.
7. have a physical disability that interferes with their ability to click a mouse button rapidly and repeatedly.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-01; Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
The Pediatric Anxiety Rating Scale (PARS) | expected average time frame of 6 weeks.
  The PARS assesses global anxiety severity across different anxiety disorders in youth.

SECONDARY OUTCOMES:
Anxiety Related Emotional Disorders - Child/Parent Version (SCARED-C/P) | expected average time frame of 6 weeks.
  The SCARED is a 41-item self and parent-report instrument designed to assess anxiety in children and adolescents.
  Screen for Child

CONTACTS AND LOCATIONS:
Locations (1):
- Tel-Aviv University, Tel Aviv, Israel